CLINICAL TRIAL: NCT02074605
Title: A Pilot Study of Neurocognitive Function in Patients Treated With Adjuvant Interferon Alpha-2b for High-Risk Melanoma
Brief Title: Cognitive Effects of Interferon in Patients With Melanoma
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Daniel Combs, Clinical Assistant, University of Arizona
Other Study IDs: 08-0389-02
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Melanoma
Keywords: Melanoma; Interferon; Cognition
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha; Introns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Observation: Patients with melanoma who qualify for interferon treatment, but choose not to receive it.
- Interferon alpha: Patients who receive high dose interferon alpha for 4 weeks
  Interventions: Biological: Interferon alpha

INTERVENTIONS:
Biological: Interferon alpha
  Other Names: Intron-A
  Groups: Interferon alpha

SUMMARY:
Interferon alpha is the only approved adjuvant biologic therapy for individuals diagnosed with high risk malignant melanoma (stage 2 or 3). There is evidence that interferon has some adverse cognitive effects on patients, but there are limited data. The investigators hypothesis is that compared to patients with melanoma who do not receive interferon, patients who have melanoma and are treated with interferon will show an objective decrease in performance on neurocognitive assessment.

This study will enroll patients with melanoma who qualify for interferon, and either decide to undergo interferon treatment or choose watchful waiting instead. All patients will be assessed with a cognitive testing battery twice. Observation patients will undergo testing at their first appointment in which they consent to the study, as well as at their next physician visit, approximately 3 months from the first visit. Interferon patients will be tested immediately prior to starting interferon, as well as immediately after completing high dose interferon.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with high risk malignant melanoma (defined as American Joint Committee on Cancer Stage IIb or greater) electing to undergo treatment with either adjuvant interferon alpha-2b, or observation only.
* Age 18 years or older.
* Karnofsky performance status greater than 60.
* Fluent English speaker.

Exclusion Criteria:

* History of neurologic or psychiatric disease that will affect patient's ability to complete protocol tests.
* Clinical or radiological evidence of brain metastasis.
* Any condition, which in the opinion of the investigator makes the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in one of these categories:
  1. Are to receive adjuvant treatment with interferon alpha-2b after complete surgical resection of high risk melanoma.
  2. Have had a complete surgical resection of high risk melanoma, but have elected not to receive interferon alpha-2b and will be observed for disease progression only.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | 1 month
  Cognitive function as assessed by a brief neurocognitive testing battery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Combs, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Result] Combs D, Baker A, Jordan S, Morgan S, Pestana L, Herring A, Jeter J, Hersh E, Cranmer LD. Screening tools for interferon-related cognitive decline in melanoma patients. J Clin Oncol 28:7s, May 2010 (suppl; abstr 8539). Abstract.
- [Result] Combs D, Baker A, Herring A, Trevor K, Jeter J, Cranmer L. Effects of high dose interferon on memory in melanoma patients. Pigment Cell and Melanoma Research 22(6):866, Dec 2009. Abstract.